CLINICAL TRIAL: NCT06586528
Title: Increasing Family Engagement in Critical Care: The NGAGE Trial (The NGAGE Trial)
Brief Title: Increasing Family Engagement in Critical Care
Acronym: NGAGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lady Davis Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Michael Goldfarb, Attending Staff, Division of Cardiology, Lady Davis Institute
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2025-4301
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-05

CONDITIONS: Family Engagement; Critical Care, Intensive Care; Patient and Family Engagement; Health Care Delivery; Family-centered Care
Keywords: Patient- and Family-Centered Care; Family Engagement; Critical Care; Intensive Care Unit; Person-Centered Care; Delivery of Health Care

STUDY DESIGN:
Intervention Model Description: In the stepped-wedge cluster design, there is random and sequential crossover of clusters from control (phase 1) to intervention (phase 2) until all clusters are exposed
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control Group: Usual Care (No Intervention): Participants in the control group will not receive access to the NGAGE tool. Participants will be able to engage in care as per current family engagement practices at each site.
- Intervention Group: Access to NGAGE Tool (Experimental): Participants in the intervention group will be provided access to the NGAGE tool.
  Interventions: Other: NGAGE tool

INTERVENTIONS:
Other: NGAGE tool — Access to NGAGE tool
  Arms: Intervention Group: Access to NGAGE Tool

SUMMARY:
The primary aim of this trial is to evaluate if the NGAGE tool improves care engagement in family members of ICU patients. The secondary objectives are to assess if the NGAGE tool improves communication, care satisfaction, psychological symptoms, and quality of life in family members of ICU patients.

The NGAGE trial is a stepped wedge cluster randomized trial of 6 Canadian adult ICUs, involving 194 family members. A family member will be considered anyone with a biological, emotional, or legal relationship with the patient and whom the patient wishes to be involved in their care. There will be random and sequential crossover of clusters from control (phase 1) to intervention (phase 2) until all clusters are exposed. The intervention group will have access to the NGAGE tool, which has modules to Learn, Engage, and Report. "Engage" allows the family member to indicate their desired engagement activity, which is then transmitted to the treating healthcare team to provide the requested activity. "Learn" contains educational capsules about the ICU environment and information about care participation. "Report" allows the family member to provide real-time feedback to the healthcare team. The primary endpoint is the FAMily Engagement (FAME) score within 1 week of ICU discharge. Secondary endpoints are family-centered outcomes, including communication quality, satisfaction, and mental health (anxiety and depression) scores within 1 week of ICU discharge, and quality of life and mental health (anxiety, depression, and post-traumatic distress symptoms) at 6 months. The mean difference of the validated FAME score, a continuous variable, will be compared between groups.

ELIGIBILITY:
Inclusion Criteria:

* Adult family members (age ≥ 18 years) of ICU patients
* Expected ICU stay ≥ 48 hours
* Able to participate in English or French

Exclusion Criteria:

* Family members who do not wish to participate in care
* Repeat admissions within the study period
* Another family member has already participated in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Estimated)
Dates: Start 2025-03-26 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
FAMily Engagement (FAME) score within 1 week of ICU discharge | 1-week post-hospital discharge
  The FAMily Engagement (FAME) tool is a self-administered 12-item questionnaire that assesses an individual's current engagement practice. FAME uses a five-point Likert scale ranging from 1 (strongly agree) to 5 (strongly disagree), and scale results are changed to a 0-100 scoring system, with higher scores indicating greater engagement in care. The following subdomains are evaluated: engagement perception, family presence, communication, education, decision-making, care contribution, and family needs. FAME includes the following engagement domains: family presence, family needs, communication and education, decision making, and direct care. FAME also captures the following family-centered care principles: dignity and respect, information sharing, participation, and collaboration.

SECONDARY OUTCOMES:
Family satisfaction in the ICU (FS-ICU) | 1-week post-hospital discharge
  The Family Satisfaction in the ICU survey (FS-ICU) is a 24-item instrument that was developed and validated to assess family satisfaction and experience with care in the ICU. Scores range from 0 to 100, with higher scores indicate greater satisfaction.
Quality of communication (QOC score) | 1-week post-hospital discharge
  The Quality of Communication tool is a 13-item questionnaire that was developed and validated in an ICU setting to measure the perceived quality of communication. Scores range from 0 to 100, with higher scores indicating better clinician-family communication.
Anxiety and depression (HADS) | 1-week post-hospital discharge
  The Hospital Anxiety and Depression Scale (HADS) is a simple to use, validated, and widely used self-reported tool to measure anxiety and depression in medical patients. The survey is composed of 14 questions: 7 depression-related and 7 anxiety-related questions. The score for each item ranges from 0 to 3, and subscale scores greater than 8 denotes anxiety or depression.
Anxiety and depression (HADS) | 6 months post-hospital discharge
  The Hospital Anxiety and Depression Scale (HADS) is a simple to use, validated, and widely used self-reported tool to measure anxiety and depression in medical patients. The survey is composed of 14 questions: 7 depression-related and 7 anxiety-related questions. The score for each item ranges from 0 to 3, and subscale scores greater than 8 denotes anxiety or depression.
Post-traumatic stress (IES-Revised) | 6 months post-hospital discharge
  The IES-Revised is a 22-item questionnaire that has been validated and is widely used for measuring post-traumatic stress symptoms and yields a total score ranging from 0 to 88 and subscale scores for the Intrusion, Avoidance, and Hyperarousal subscales. Items are rated on a 5-point scale ranging from 0 (not at all) to 4 (extremely). High scores indicate greater severity of PTSD.
Quality of life (EuroQOL-5D-5L score) | 6 months post-hospital discharge
  The EuroQOL-5D-5L is a 5-item questionnaire that has been validated and is widely used for measuring health-related quality of life. Each dimension has five response levels: no problems (Level 1); slight; moderate; severe; and extreme problems (Level 5). The scores are combined to generate a single index value for overall health status. EQ-5D-5L index scores range from -0.59 to 1, where 1 is the best possible health state

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Goldfarb, MD, MSc, Principal Investigator — Lady Davis Institute, McGill University, Jewish General Hospital
Locations (2):
- Canada (2):
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No